CLINICAL TRIAL: NCT03639948
Title: Neoadjuvant Phase II Study of Pembrolizumab And Carboplatin Plus Docetaxel in Triple Negative Breast Cancer
Acronym: NeoPACT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-NeoPACT
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Triple-negative Breast Cancer
Keywords: Pembrolizumab; Carboplatin; Docetaxel; Pegfilgrastim; breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Carboplatin; Docetaxel; pembrolizumab; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Carboplatin & Docetaxel plus Pembroluzimab (Experimental): Carboplatin (Area under the curve [AUC] 6 intravenously [IV]) and Docetaxel (75 milligrams per meter squared [mg/m2], IV) plus Pembrolizumab (200 milligrams [mg], IV) every 21 days for 6 cycles.
  Pegfilgrastim 6 mg subcutaneous (SC) Day 2 of each cycle.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Drug: Pembrolizumab; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Carboplatin — Intravenous solution
Drug: Docetaxel — Intravenous solution
Drug: Pembrolizumab — Intravenous solution
Drug: Pegfilgrastim — Injectable product

SUMMARY:
The standard treatment for women with stage I, II, and III triple-negative breast cancer (TNBC) includes chemotherapy and surgery, with or without radiation therapy. However, because TNBC is usually more aggressive, harder to treat, and more likely to come back, it is associated with poor long-term outcomes (survival rates) when compared to other types of breast cancer. Therefore, researchers are studying how new drugs and treatment combinations can improve the outcome of patients with TNBC. This study will test effectiveness of immune therapy (Pembrolizumab is an "immunotherapy" that is expected to work with the body's immune system to help fight cancer) in combination with chemotherapy given before surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of participant to understand this study, and participant willingness to sign a written informed consent for this trial.
* Histologically confirmed stage I , II or III TNBC (triple-negative breast cancer).
* No previous definitive ipsilateral breast surgery for the current breast cancer.
* No previous chemotherapy, endocrine therapy, or radiation therapy with therapeutic intent for this cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Adequate cardiac function
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP)
  * A WOCBP who agrees to follow contraceptive guidelines.

Key Exclusion Criteria:

* Current or anticipated use of other investigational agents while participating in this study.
* Participant has received chemotherapy, radiotherapy, or surgery for the treatment of breast cancer.
* Participant has metastatic disease.
* Participant has inflammatory breast cancer.
* Participants with concomitant or previous malignancies within the last 5 years are excluded from the study.

  * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. ductal carcinoma in situ (DCIS), carcinoma in situ of the cervix) that have undergone potential curative therapy are not excluded.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to agents used in this study.
* Participant has received prior therapy with an anti-programmed death (PD) -1, anti-PD-ligand (L)-1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory thymus lymphocyte (T-cell) receptor.
* Subject has received a live vaccine within 30 days prior to the first dose of study drug.
* Participant is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Participant has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of Pembrolizumab.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has a history of (non-infectious) pneumonitis that required steroids, or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B or known active Hepatitis C virus.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects
Enrollment: 120 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2024-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Sharma, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (9):
- United States (9):
  - The University of Kansas Cancer Center (KUCC), Fairway, Kansas
  - The University of Kansas Cancer Center, West Clinic, Kansas City, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center, Overland Park Clinic, Overland Park, Kansas
  - The University of Kansas Cancer Center, North Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center, Lee's Summit Clinic, Lee's Summit, Missouri
  - The University of Kansas Medical Center, North Kansas City, Missouri
  - Texas Oncology- Baylor, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma P, Stecklein SR, Yoder R, Staley JM, Schwensen K, O'Dea A, Nye L, Satelli D, Crane G, Madan R, O'Neil MF, Wagner J, Larson KE, Balanoff C, Kilgore L, Phadnis MA, Godwin AK, Salgado R, Khan QJ, O'Shaughnessy J. Clinical and Biomarker Findings of Neoadjuvant Pembrolizumab and Carboplatin Plus Docetaxel in Triple-Negative Breast Cancer: NeoPACT Phase 2 Clinical Trial. JAMA Oncol. 2024 Feb 1;10(2):227-235. doi: 10.1001/jamaoncol.2023.5033. PMID 37991778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 patients were found to be ineligible after enrollment and are not included in assessment for study outcomes.
Groups:
- Experimental: Carboplatin & Docetaxel Plus Pembrolizumab: Carboplatin (Area under the curve [AUC] 6 intravenously [IV]) and Docetaxel (75 milligrams per meter squared [mg/m2], IV) plus Pembrolizumab (200 milligrams [mg], IV) every 21 days for 6 cycles.
  Pegfilgrastim 6 mg subcutaneous (SC) Day 2 of each cycle.
  Carboplatin: Intravenous solution
  Docetaxel: Intravenous solution
  Pembrolizumab: Intravenous solution
  Pegfilgrastim: Injectable product
Period: Overall Study
Arm/Group | Experimental: Carboplatin & Docetaxel Plus Pembrolizumab
Started | 115
Completed | 115
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Experimental: Carboplatin & Docetaxel Plus Pembroluzimab: Carboplatin (Area under the curve [AUC] 6 intravenously [IV]) and Docetaxel (75 milligrams per meter squared [mg/m2], IV) plus Pembrolizumab (200 milligrams [mg], IV) every 21 days for 6 cycles.
  Pegfilgrastim 6 mg subcutaneous (SC) Day 2 of each cycle.
  Carboplatin: Intravenous solution
  Docetaxel: Intravenous solution
  Pembrolizumab: Intravenous solution
  Pegfilgrastim: Injectable product
Arm/Group | Experimental: Carboplatin & Docetaxel Plus Pembroluzimab
Number analyzed (Participants) | 115
Age, Continuous [Median (Full Range); unit: years] | 50 [27 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 112
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 91
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 115
Lymph node status [Count of Participants; unit: Participants]
  Negative | 70
  Positive | 45
T stage [Count of Participants; unit: Participants] — Measure Description: Primary tumor stage, as defined by the 8th edition of the American Joint Committee on Cancer's staging manual. T stage indicates the size or extent of the primary tumor. T1: tumor ≤20 mm in greatest dimension; T2:tumor >20 mm but ≤50 mm in greatest dimension; T3: tumor >50 mm in greatest dimension; T4: tumor of any size with direct extension to the chest wall and/or to the skin (ulceration or skin nodules).
  Participants
    T1 | 21
    T2 | 73
    T3 | 21
    T4 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: Defined as the percentage of patients with PCR, as evidenced by absence of invasive disease in breast and axillary lymph nodes determined by histopathological examination.
Time Frame: Up to 25 weeks
Population: Evaluable for pathologic response
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Carboplatin & Docetaxel Plus Pembroluzimab
Number analyzed (Participants) | 111
Participants | 64

2. Secondary Outcome: Minimal Residual Disease (MRD) Rate
Description: Defined as the percentage of patients with MRD, as evidenced by residual cancer burden (RCB) score of 0/1. Residual cancer burden score for each patient is calculated using surgical pathology parameters using an online tool (http://www3.mdanderson.org/app/medcalc/index.cfm?pagename=jsconvert3).
Time Frame: Up to 25 weeks
Population: Residual cancer burden (RCB) class available
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Carboplatin & Docetaxel Plus Pembroluzimab
Number analyzed (Participants) | 110
Participants | 76

3. Secondary Outcome: Percentage of Participants With Event-free Survival (EFS) as Assessed by Kaplan-Meier Method
Description: Percentage of patients with EFS as assessed by Kaplan-Meier method. EFS is defined as time from diagnosis to first invasive locoregional or distant recurrence, study treatment-related death, or breast cancer-related death
Time Frame: Up to 3 years
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: Survival percentage by Kaplan-Meier
Arm/Group | Experimental: Carboplatin & Docetaxel Plus Pembroluzimab
Number analyzed (Participants) | 115
Survival percentage by Kaplan-Meier | 86 [77 to 95]

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Adverse events occurring in 5% or more of participants in the intent-to-treat population. Patients were systematically evaluated for toxicity at each visit. Per protocol, only adverse events determined to be definitely related/probably related/possibly related to study treatment, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, are to be reported.
Arm/Group | Experimental: Carboplatin & Docetaxel Plus Pembroluzimab
All-Cause Mortality (participants affected / at risk) | 11/115
Serious Adverse Events (participants affected / at risk) | 17/115
Other Adverse Events (participants affected / at risk) | 115/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Carboplatin & Docetaxel Plus Pembroluzimab (N=115)
Colitis (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Osteomyelitis (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 1
Cellulitis (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Fever (General disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Flu-like symptoms (General disorders) | 1
Bacteremia (Infections and infestations) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Creatinine increased (Investigations) | 1
Enteritis (Gastrointestinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Carboplatin & Docetaxel Plus Pembroluzimab (N=115)
Fatigue (General disorders) | 87
Diarrhea (Gastrointestinal disorders) | 72
Nausea (Gastrointestinal disorders) | 68
Peripheral sensory neuropathy (Nervous system disorders) | 47
Constipation (Gastrointestinal disorders) | 44
Dysgeusia (Nervous system disorders) | 41
Alopecia (Skin and subcutaneous tissue disorders) | 39
Mucositis oral (Gastrointestinal disorders) | 39
Arthralgia (Musculoskeletal and connective tissue disorders) | 32
Rash (Skin and subcutaneous tissue disorders) | 28
Watering eyes (Eye disorders) | 27
Anorexia (Metabolism and nutrition disorders) | 26
Edema limbs (General disorders) | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 24
Anemia (Blood and lymphatic system disorders) | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 20
Nail discoloration (Skin and subcutaneous tissue disorders) | 20
Insomnia (Psychiatric disorders) | 19
Headache (Nervous system disorders) | 16
Hot flashes (Vascular disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13
Fever (General disorders) | 13
Hypomagnesemia (Investigations) | 13
Dehydration (Metabolism and nutrition disorders) | 12
Vomiting (Gastrointestinal disorders) | 12
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10
Hypokalemia (Investigations) | 10
Dizziness (General disorders) | 9
Dermatitis (Skin and subcutaneous tissue disorders) | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9
Creatinine increased (Investigations) | 6
Abdominal pain (Gastrointestinal disorders) | 6
Platelet count decreased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03639948/Prot_SAP_000.pdf